CLINICAL TRIAL: NCT00593034
Title: Medical Office Intervention for Adolescent Drug Use - Research Supplement for Under-represented Minorities
Brief Title: Medical Office Intervention for Adolescent Drug Use - Attention Study Supplement
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: John R. Knight, MD, Children's Hospital Boston
Other Study IDs: R01DA014553-03S1 (NIH)
Record Dates: First submitted 2008-01-03; First posted 2008-01-14 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Substance-related Disorders
Keywords: Alcohol abuse; Drug abuse
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Participants in this study will be 12-21 year old patients who have been referred to the Adolescent Substance Abuse Program for evaluation of drug or alcohol use and are participating in the parent study, "Medical Office Intervention for Adolescent Drug Abuse."

SUMMARY:
This study will use the CCPT II to assess attention in 12-21 year olds enrolled in a randomized controlled trial of a brief behavioral treatment for substance abuse.

This study will describe at baseline levels of attention using a well validated instrument (Connors Continuous Performance Test II) and explore the association between attention levels and substance use. The primary study hypothesis is that lower initial levels of substance use (as measured by percent days abstinent) will be associated with higher attention levels. We envision that this data will inform a better understanding of how attention may modify treatment response.

DETAILED DESCRIPTION:
Research among adolescents with substance use problems presents unique challenges to investigators. Issues with recruitment, confidentiality, and follow-up have been cited as common limitations to research in this area. One likely contributor to decreased treatment persistence and follow-up is the limited ability to sustain attention that many adolescents, especially those with substance problems, may manifest. (Taper, 2002) Thus, assessing attention before beginning substance abuse treatment has the potential not only to inform the science of adolescent addiction medicine, but also to guide the development of therapies to specifically address attention deficits among adolescent substance users. Adolescent outpatients being treated for substance problems have not been systematically studied for clinical or subclinical attention levels.

The primary aims this study are as follows:

1. To test the feasibility of administering the Connors Continuous Performance Test II (CCPT II), a well validated measure of attention, to a sample of 12-21 year old patients receiving treatment for substance abuse.
2. To obtain baseline descriptive statistics on the CCPT II in a previously understudied group of young patients receiving treatment for substance abuse.
3. To estimate the magnitude of the association between substance use and levels of attention at baseline before treatment.
4. To explore the degree to which attention may affect response to substance abuse treatment in general and specifically motivational interviewing.

ELIGIBILITY:
Inclusion Criteria:

* CRAFFT score of 1 or more
* Have used cannabis, alcohol or another drug on at least two occasions during the 30 days preceding their visit
* Can read and understand English

Exclusion Criteria:

* Require immediate hospitalization or referral to residential substance abuse treatment
* Will not be available to complete the study assessments over the next 9 months.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants in this study will be 12-21 year old patients who have been referred to the Adolescent Substance Abuse Program for evaluation of drug or alcohol use and are participating in the parent study, "Medical Office Intervention for Adolescent Drug Abuse."
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Score on the Connors Continuous Performance Test II (CCPT II) | Baseline

SECONDARY OUTCOMES:
Percentage of days abstinent | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Knight JR, Shrier LA, Bravender TD, Farrell M, Vander Bilt J, Shaffer HJ. A new brief screen for adolescent substance abuse. Arch Pediatr Adolesc Med. 1999 Jun;153(6):591-6. doi: 10.1001/archpedi.153.6.591. PMID 10357299
- [Background] Knight JR, Sherritt L, Shrier LA, Harris SK, Chang G. Validity of the CRAFFT substance abuse screening test among adolescent clinic patients. Arch Pediatr Adolesc Med. 2002 Jun;156(6):607-14. doi: 10.1001/archpedi.156.6.607. PMID 12038895
- See also: Web site for the Center for Adolescent Substance Abuse Research, parent research group for the project. — http://www.ceasar.org